CLINICAL TRIAL: NCT06578780
Title: Design and Delivery Preferences for Exercise Intervention in People With Spinal Cord Injury: a Pilot Discrete Choice Experiment
Brief Title: Design and Delivery Preferences for Exercise Intervention in People With Spinal Cord Injury
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Yumi Kim, Scientist I, University of Alabama at Birmingham
Other Study IDs: 300012355; 1143477 (Other Grant/Funding Number: Craig H. Neilsen Foundation)
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injury; Exercise; Adults
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research study aims to explore people's understanding of physical activity behavior and perceptions of what a physical activity program should include for supporting initiation and continuous participation. This study will enroll up to 30 adults (18 or over) with spinal cord injury. The study will use a discrete choice experiment (DCE) design that implements both quantitative (development of preference survey) and qualitative approaches (systematic review; test of preference survey).

DETAILED DESCRIPTION:
Aim 1. To explore individual preferences and needs that are related to engaging in a physical activity behavior using both qualitative and quantitative approaches.

The identification of attributes will be achieved through (a) qualitative interviews of 30 adults living with SCI, (b) expert opinion of 10 healthcare professionals who have at least 5 years of work experience with SCI patients and in the field of SCI research, and (c) a rapid review of literature reporting on preferred design, equipment, and/or delivery methods for physical activity/exercise programs for people with SCI. For the qualitative approach, we will use semi-structured, one-on-one interviews. Using deductive content analysis, we will generate participant-informed categories that aligned with the "what, when, where, and who" of exercise programs for people with SCI to develop an initial DCE survey.

Participants who take part in this study will engage in two one-on-one interviews that last approximately 1 hour each, depending on how much information is shared with the researcher. The interview will be conducted by the lead researcher via phone or video conference call. The interview will be audio-recorded, which will later be transcribed. The interview will ask questions about your interests, preferences, and wants for a physical activity program that supports initiation and long-term participation. The information shared during the interview will be used to create a preference survey, and the interviewed participants will be contacted again to complete the developed survey and a second interview to see whether the survey fully covered the choices of their needs and wants.

Aim 2. To develop and refine a quantitative DCE survey that contains essential attributes and preference levels for physical activity participation.

The developed initial DCE from Aim 1 will be further refined through the survey responses and feedback from the interviewed participants with SCI as well as iterative discussions with the interviewed healthcare professionals. The evaluation criteria will follow the DCE design guidelines, such as the clarity of the attributes, attribute descriptions, and preference levels; redundancy of attributes and levels defined; and level of burden.

Aim 3. 3-1. To examine which attributes and preference levels are essential and more likely to be accepted for increasing participation in a physical activity intervention.

The developed and refined DCE from Aim 1 and 2 will be pilot tested among 100 people with SCI, who were not involved in the qualitative interview and survey refinement processes. Using conjoint analysis techniques, we will develop prediction models based on the possible combinations of attributes and levels (e.g., 24 combinations = 3 levels of "what" x 2 of "when" x 2 of "where" x 2 of "who").

3-2. To examine whether these preferences vary by participants' personal and clinical characteristics, such as age, functional level, residential area (urban vs. rural), and self-reported physical activity and motivational readiness to physical activity behavior change (pre-intenders, intenders, actors).

Hypothesis:

Adults with SCI who are currently meeting/exceeding physical activity guidelines (actors) will choose a self-guided physical activity program over a supervised, instructor-led program. Adults with SCI who have a high level of self-regulatory skills (goal setting and planning) will choose a self-guided physical activity program over a supervised, instructor-led program.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years) with spinal cord injury
* able to converse and read in English

Exclusion Criteria:

* presence of cognitive impairment that prevents adhering to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adults with spinal cord injury interested in participating in this study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Demographics & clinical information | Baseline, during the first interview
  age, ethnicity, race, date of spinal cord injury onset, injury level, injury type
Physical activity | Baseline, during the first interview
  Complete LTPAQ-SCI online survey (mins of physical activity per week)
Physical activity | 3-month follow-up, before the second interview
  Complete LTPAQ-SCI online survey (mins of physical activity per week)
Preference survey | 3-month follow-up, before the second interview
  Developed preference survey based on the first interview

CONTACTS AND LOCATIONS:
Overall Officials: Yumi Kim, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Wellness, Health and Research Facility (WHARF), Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No